CLINICAL TRIAL: NCT02962648
Title: An Open-label, Multicentre, Extension Trial to Assess the Safety of Re-dosing of Intravenous Iron Isomaltoside/Ferric Derisomaltose (Monofer®/Monoferric®)
Brief Title: An Extension Trial to Assess the Safety of Re-dosing of Iron Isomaltoside/Ferric Derisomaltose (Monofer®/Monoferric®)
Acronym: FERWON-EXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IDA/CKD-EXT-01
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-01

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency Anaemia
Keywords: Iron Deficiency Anemia; Iron Deficiency Anaemia; IDA; Intravenous iron replacement therapy; Chronic Kidney Disease; CKD; Iron isomaltoside; Ferric derisomaltose; Monofer; Monoferric; Monover; Monofar; Monoferro
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — iron isomaltoside 1000; ferric derisomaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iron isomaltoside/ferric derisomaltose (Experimental): Administered IV
  Interventions: Drug: Iron isomaltoside/ferric derisomaltose

INTERVENTIONS:
Drug: Iron isomaltoside/ferric derisomaltose — Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  The dose of iron isomaltoside/ferric derisomaltose for the individual subject was set to 1000 mg. The dose was diluted in 100 mL 0.9 % sodium chloride from the site's supply and administered over approximately 20 minutes using IV infusion.
  Other Names: Monofer®, Monoferric®, Monover®, Monofar®, Monoferro®

SUMMARY:
Evaluate safety and efficacy of intravenous (IV) iron isomaltoside/ferric derisomaltose re-dosing, in subjects who were previously treated with iron isomaltoside/ferric derisomaltose.

DETAILED DESCRIPTION:
Among the various formulations of parenteral iron that are currently available, iron isomaltoside/ferric derisomaltose may allow flexibility in terms of high and rapid dosing. Up to now, most clinical trials with intravenous (IV) iron treatment were of 4-12 weeks in duration; longer trials are warranted to follow-up on long-term safety.

The aim of the trial was to evaluate the safety and efficacy of IV iron isomaltoside/ferric derisomaltose re-dosing in subjects who were previously treated with iron isomaltoside/ferric derisomaltose in lead-in trials.

This was a 6-months extension trial lasting 26 weeks. Eligible subjects attended 5 visits: screening, baseline (subjects treated with a single IV dose of 1000 mg iron isomaltoside/ferric derisomaltose), and follow-up visits at week 2, 13, and 26 weeks after the IV dose, for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Completed one of the lead-in trials
2. Randomised and dosed with iron isomaltoside/ferric derisomaltose in one of the lead-in trials.
3. Haemoglobin (Hb) of ≤ 11 g/dL
4. Screening serum ferritin (s-ferritin) ≤ 100 ng/mL, or ≤ 300 ng/mL if transferrin saturation (TSAT) ≤ 30 %
5. Willingness to participate and signing the informed consent form (ICF)

Exclusion Criteria:

1. Intravenous (IV) iron treatment between the lead-in trial and screening
2. During 30-day period prior to screening or during the trial period; has or will be treated with a red blood cell transfusion, radiotherapy, and/or chemotherapy
3. Received an investigational drug within 30 days of screening
4. Decompensated liver cirrhosis or active hepatitis
5. Pregnant or nursing women.
6. Any other laboratory abnormality, medical condition, or psychiatric disorders which, in the opinion of the Investigator, will put the subject's disease management at risk or may result in the subject being unable to comply with the trial requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S Clinical and Non-clinical Research, Study Director — Pharmacosmos A/S
Locations (20):
- United States (20):
  - Pharmacosmos Investigational Site, Chula Vista, California
  - Pharmacosmos Investigational Site 1, La Mesa, California
  - Pharmacosmos Investigational Site 2, La Mesa, California
  - Pharmacosmos Investigational Site, Northridge, California
  - Pharmacosmos Investigational Site, Porterville, California
  - Pharmacosmos Investigational Site, Doral, Florida
  - Pharmacosmos Investigational Site, Hialeah, Florida
  - Pharmacosmos Investigational Site, Miami, Florida
  - Pharmacosmos Investigational Site, Miami Lakes, Florida
  - Pharmacosmos Investigational Site, West Palm Beach, Florida
  - Pharmacosmos Investigational Site, Baton Rouge, Louisiana
  - Pharmacosmos Investigational Site, Metairie, Louisiana
  - Pharmacosmos Investigational Site, New Orleans, Louisiana
  - Pharmacosmos Investigational Site, Shreveport, Louisiana
  - Pharmacosmos Investigational Site, Plainsboro, New Jersey
  - Pharmacosmos Investigational Site, Albuquerque, New Mexico
  - Pharmacosmos Investigational Site, Chattanooga, Tennessee
  - Pharmacosmos Investigational Site, Houston, Texas
  - Pharmacosmos Investigational Site 1, San Antonio, Texas
  - Pharmacosmos Investigational Site 2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 193 subjects were screened and 103 subjects were enrolled into the trial.
Pre-assignment Details: Subjects enrolled in this extension trial had previously participated in the lead-in trials IDA-03 (52%, NCT02940886), CKD-04 (32%, NCT02940860), and IDA-01 (16%, NCT02130063).
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  Subjects received iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) as a single IV infusion of 1000 mg at the baseline visit.
Period: Overall Study
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Started | 103
Completed | 94
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Subject had problems with transportation | 2

BASELINE CHARACTERISTICS:
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose, administered IV
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (15.7)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 82
  65-84 years | 18
  >84 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 103
Current smoker [Count of Participants; unit: Participants]
  Yes | 8
  No | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Drug Reactions (ADR)
Description: Safety
  Evaluate the number of subjects with adverse drug reactions (ADRs), defined as AEs that were assessed by the investigator as related or possible related to the investigational product.
Time Frame: Baseline to week 26
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 102
Participants | 5

2. Secondary Outcome: Incidence of Protocol-defined Serious or Severe Hypersensitivity Reactions
Description: Safety.
  For this endpoint, the number of participants with serious or severe hypersensitivity reactions were evaluated. The hypersensitivity terms that were included in the analysis were those that started or after the first dose of treatment (i.e. treatment emergent). The terms used to define hypersensitivity were those specified by the Standardised MedDRA Queries (SMQ) for hypersensitivity, plus four additional terms: Loss of consciousness; Seizure; Syncope; Unresponsiveness.
  The potential hypersensitivity AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  Results show only those participants that had adjudicated and confirmed serious or severe hypersensitivity reactions.
Time Frame: Baseline to week 26
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 102
Participants | 0

3. Secondary Outcome: Composite Cardiovascular Adverse Events (AEs)
Description: Safety
  Results show the composite cardiovascular AEs, that started on or after the first dose of treatment (i.e. treatment emergent) up to month 6.
  The reported potential cardiovascular AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  The potential cardiovascular AEs included the following:
  * Death due to any cause
  * Non-fatal myocardial infarction
  * Non-fatal stroke
  * Unstable angina requiring hospitalisation
  * Congestive heart failure requiring hospitalisation or medical intervention
  * Arrhythmias
  * Hypertension
  * Hypotension
  Results show only those participants that had adjudicated and confirmed treatment-emergent composite cardiovascular AEs.
Time Frame: Baseline to week 26
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 102
Participants | 6

4. Secondary Outcome: Time to First Composite Cardiovascular Safety AE
Description: Safety
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit. Only the adjudicated and confirmed composite cardiovascular safety AEs, as judged by the Clinical Endpoint Adjudication Committee (CEAC), were considered for this endpoint.
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit.
Time Frame: Baseline, week 2, 13, and 26
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Median (95% Confidence Interval); unit: week
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 102
week | NA [NA to NA] — The number of adjudicated and confirmed composite cardiovascular safety AEs was too low (N=6) for estimation of median and 95 % CI.

5. Secondary Outcome: S-phosphate <2 mg/dL at Any Time From Baseline to Week 26
Description: Safety
  Results show the number of trial participants and their status of s-phosphate <2 mg/dL, at any time from baseline to week 26.
Time Frame: Baseline to week 26
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 102
Participants
  Yes | 8
  No | 94

6. Secondary Outcome: Change in Hb From Baseline to Week 2, 13, and 26
Description: Efficacy.
  Change in Hb from baseline to week 2, 13, and 26.
Time Frame: Baseline, week 2, 13, and 26
Population: Intention-to-treat (ITT) analysis set: included all subjects, except for screening failures and subjects withdrawn before visit 2 (baseline).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 103
g/dL
  Week 2: number analyzed (Participants) | 100
  Week 2 | 1.23 (1.40)
  Week 13: number analyzed (Participants) | 97
  Week 13 | 1.73 (1.83)
  Week 26: number analyzed (Participants) | 93
  Week 26 | 1.34 (1.93)

7. Secondary Outcome: Change in S-ferritin From Baseline to Week 2, 13, and 26
Description: Efficacy.
  Change in s-ferritin from baseline to week 2, 13, and 26.
Time Frame: Baseline, week 2, 13, and 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 103
ng/mL
  Week 2: number analyzed (Participants) | 100
  Week 2 | 255.6 (177.9)
  Week 13: number analyzed (Participants) | 98
  Week 13 | 87.9 (123.6)
  Week 26: number analyzed (Participants) | 94
  Week 26 | 93.9 (180.4)

8. Secondary Outcome: Change in Transferrin Saturation (TSAT) From Baseline to Week 2, 13, and 26
Description: Efficacy
  Change in transferrin saturation (TSAT) from baseline to week 2, 13, and 26.
  TSAT is the value of serum iron divided by the total iron-binding capacity and the unit is %, which referrers to % of iron-binding sites of transferrin being occupied by iron.
Time Frame: Baseline, week 2, 13, and 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 103
percentage of saturation
  Week 2: number analyzed (Participants) | 100
  Week 2 | 8.16 (11.87)
  Week 13: number analyzed (Participants) | 98
  Week 13 | 4.42 (10.81)
  Week 26: number analyzed (Participants) | 94
  Week 26 | 1.78 (10.63)

9. Secondary Outcome: Change in S-iron From Baseline to Week 2, 13, and 26
Description: Efficacy.
  Change in s-iron from baseline to week 2, 13, and 26.
Time Frame: Baseline, week 2, 13, and 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
Number analyzed (Participants) | 103
μg/dL
  Week 2: number analyzed (Participants) | 98
  Week 2 | 21.1 (50.5)
  Week 13: number analyzed (Participants) | 96
  Week 13 | 10.7 (45.4)
  Week 26: number analyzed (Participants) | 92
  Week 26 | 4.0 (44.1)

ADVERSE EVENTS:
Time Frame: From the time subjects signed the informed consent form (CRF) until they completed the trial, all adverse events (AEs) or serious adverse events (SAEs) were recorded in the CRF. The actual study duration was 6 months (or shorted if the trial was discontinued). Overall, eligible subjects participated in the trial for approximately 6.5 months (including a 14-day screening period).
Description: An AE was described as follows: the nature of the event was described in precise, standard medical terminology (i.e. not necessarily the exact words used by the subject). If known, a specific diagnosis was stated. Furthermore, the Investigator described an AE regarding seriousness, severity, relatedness, and outcome.
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose
All-Cause Mortality (participants affected / at risk) | 1/193
Serious Adverse Events (participants affected / at risk) | 13/102
Other Adverse Events (participants affected / at risk) | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=102)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Endometritis (Infections and infestations) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=102)
Fatigue (General disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the study results. Before submission for publication or presentation, Institution shall allow Sponsor not less than 90 days to review any manuscript and not less than 30 days to review any poster presentation, abstract, or any other written or oral material which describes or discloses the study results. If sponsor so requests in writing, Institution shall withhold any publication or presentation for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT02962648/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02962648/SAP_001.pdf